CLINICAL TRIAL: NCT02272400
Title: Image Guided Radiotherapy (IGRT) for Prone Partial Breast Irradiation (PBI)
Brief Title: Image Guided Radiotherapy (IGRT) for Prone Partial Breast Irradiation
Acronym: PBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-582
Record Dates: First submitted 2014-10-08; First posted 2014-10-23 (Estimated); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer
Keywords: image guided radiation therapy; partial breast irradiation; breast cancer; breast; cancer; breast preservation; IGRT; PBI
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — Radiotherapy, Image-Guided

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IGRT of prone partial breast (Experimental): IGRT for prone partial breast irradiation (PBI): All patients will be treated prone with 6 Gy/fraction delivered in 5 fractions over a 1-week period for a total dose of 30 Gy.
  Interventions: Other: IGRT for prone partial breast irradiation (PBI)

INTERVENTIONS:
Other: IGRT for prone partial breast irradiation (PBI) — IGRT for prone partial breast irradiation (PBI): All patients will be treated prone with 6 Gy/fraction delivered in 5 fractions over a 1-week period for a total dose of 30 Gy. Simulation and treatment will be started within 50 days from surgery in order to maximize the chances of optimal lumpectomy cavity visualization on the planning and cone beam CT scans. All patients will be followed monthly for the first 90 days then q3 months for the first year, then yearly for the next 10 years.
  Other Names: IGRT; PBI

SUMMARY:
Partial breast irradiation (PBI) is becoming a new paradigm for breast cancer radiation.[1] No type I or II evidence is currently available to demonstrate equivalence to standard whole breast radiotherapy, and a prospective randomized trial jointly sponsored by NSABP and RTOG (NSABP B-39 and RTOG 0413) is currently accruing patients, comparing whole breast radiotherapy to PBI, either by brachytherapy or external beam techniques (EB). Until the results of this or similar trials are available, PBI remains a research domain, and it should be offered to patients only in the context of a clinical experimental protocol.

DETAILED DESCRIPTION:
Despite the fact that less extensive experience than that of brachytherapy is available, PBI delivery through an external-beam has many advantages. First of all, it is likely to be more acceptable to the patient since it is non-invasive and it does not require a surgical procedure or anesthesia. Moreover, since it is delivered after surgery, the pathological analysis of the segmental mastectomy specimen is available to inform the selection of the best candidates. In addition, EB-PBI is likely to become more widely reproducible, since it does not rely on the experience and skills of the radiation oncologist performing the brachytherapy implant. Besides, once the technique is established, it can be widely applied at any facility provided with a linear accelerator, without the risk presented by some brachytherapy approaches that can not be completed because of the unfavorable interplay of patient's anatomy with the technical limitations of the applicator. Finally, in terms of health care economics, an external beam approach spares the costs of an extra surgical procedure and that of several days of hospitalization (in the case of LDR brachytherapy).

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women defined as either:

  1. at least 2 years without menstrual period or
  2. patients older than 50 with serological evidence of post-menopausal status or
  3. hysterectomized patients of any age with FSH confirmation of post-menopausal status
* pT1 breast cancer, excised with negative margins
* pN0 or sentinel node negative or N0 clinically if the tumor is < 1 cm in size

Exclusion Criteria:

* Previous radiation therapy to the ipsilateral breast
* Presence of a proportion of DCIS in the core biopsy specimen which is compatible with extensive intraductal component (EIC)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2007-08-07 (Actual); Primary Completion 2014-10-29 (Actual); Study Completion 2014-10-29 (Actual)

PRIMARY OUTCOMES:
Measure the outcome of applying IGRT to PBI | 10 years
  Apply IGRT to PBI as part of breast preservation in post-menopausal women with T1 breast cancers and acquire preliminary data on the role of this tool to assure correct targeting.
  Measure local recurrence within the field of conformal radiation as well as local recurrence outside the field

SECONDARY OUTCOMES:
Feasibility of accelerated dose fractionation | 1 - 10 years
  Assess the feasibility of an accelerated dose fractionation (600 cGy x 5) when given over five consecutive day by measuring the acute and late radiation toxicity
Genetic pre-disposition of patient to post-treatment radiation fibrosis | 1 - 10 years
  Prospectively determine if genetic factors can be identified which may predispose a patient to the development of post-treatment radiation fibrosis

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Perez, M.D., Principal Investigator — NYU Langone Medical Center
Locations (1):
- Laura and Isaac Perlmutter Cancer Center at NYU, New York, New York, United States